CLINICAL TRIAL: NCT03247972
Title: Antiplatelet Effects of Evolocumab in Patients With Peripheral Arterial Disease
Status: Terminated | Type: Observational
Why Stopped: Research group transferred to another hospital
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2584
Record Dates: First submitted 2017-06-29; First posted 2017-08-14 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-06

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — evolocumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with peripheral artery disease receiving evolocumab + high dose statins: Adult patients with a history of Peripheral Artery Disease (PAD) defined as one or more of the following:
  * Documented history of PAD
  * Previous limb or foot amputation for arterial vascular disease (i.e., excludes trauma),
  * Carotid artery disease (defined as >50% stenosis or prior revascularization )
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — Sixty subjects will be treated with high dose statins for 8 weeks followed by 8 weeks of high dose statin + evolocumab (420mg/4 wk) therapy.

SUMMARY:
This investigation will be conducted in subjects >18 years of age with PAD. Platelet activation and aggregation, and biomarkers associated with platelet activation, oxidative stress, and inflammation will be assessed prior to initiation of study-HD statin therapy (baseline), after 8 weeks of high-dose statins and 24 hours and 8 weeks after high dose statin + evolocumab therapy

DETAILED DESCRIPTION:
Monoclonal antibodies against PCSK9 are innovative agents that provide very potent LDL reduction when administered on top of statins. PCSK9 antibodies prevent LDL receptor degradation and enhance circulatory LDL cholesterol clearance. High LDL is a major risk factor for PAD and therefore lipid-lowering therapy constitutes another important therapeutic intervention for patients with PAD. Evolocumab is a common PCSK-9 inhibitor that has been shown to reduce plasma LDL. In this study sixty subjects will be treated with high dose statins for 8 weeks followed by 8 weeks of high dose statin + evolocumab (420mg/4 wk) therapy to determine the effect of Repatha on markers of cholesterol, thrombosis, and inflammation.

ELIGIBILITY:
Criteria: Inclusion Criteria:

Symptomatic PAD, as evidenced by either

* intermittent claudication with ABI <0.90, or
* peripheral arterial revascularization procedure, or
* amputation due to atherosclerotic disease.
* Subject may be of either sex and of any race, and must be >18 years of age.
* Subject agrees to not participate in any other investigational or invasive clinical study for a period of 4 months during the study period
* Subject must be willing and able to give appropriate informed consent.
* The subject is able to read and has signed and dated the informed consent document including authorization permitting release of personal health information approved by the investigator's Institutional Review Board (IRB).

Exclusion Criteria:

* Prior use of any PCSK9 inhibition treatment Participation in any investigational study within the last 60 days.
* Severe renal dysfunction, defined as an eGFR <20 mL/min/1.73 m2 at screening
* Active liver disease or hepatic dysfunction, defined as AST or ALT >3 x ULN as determined by central laboratory analysis at screening
* Recipient of any major organ transplant (e.g., lung, liver, heart, bone marrow, renal)
* Known major active infection or major hematologic, renal, metabolic, gastrointestinal, or endocrine dysfunction in the judgment of the investigator
* Malignancy (except non-melanoma skin cancers, cervical in situ carcinoma, breast ductal carcinoma in situ, or stage 1 prostate carcinoma) within the last 10 years
* Subject has received drugs via a systemic route that have known major interactions with background statin therapy within 1 month before randomization or is likely to require such treatment during the study period (e.g. cyclosporine, clarithromycin, HIV protease inhibitors, gemfibrozil)
* Female subject who is unwilling to use at least 2 effective birth control methods for at least 1 month before screening and 15 weeks after the end of treatment with investigational products, unless the subject is sterilized or postmenopausal.
* Subject is pregnant or breast feeding, or planning to become pregnant or to breastfeed during receipt of investigational products and within 15 weeks after the end of study treatment
* Known previous hypersensitivity reaction/s to the investigational products' active components and excipients.
* Subjects treated with any antithrombotic agents except aspirin.
* Subject likely to not be available to complete all protocol-required study visits or procedures, to the best of the subject's and investigator's knowledge
* History or evidence of any other clinically significant disorder, condition, or disease other than those outlined above that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty patients with symptomatic PAD, as evidenced by:
  * either intermittent claudication with ABI <0.90, or
  * peripheral arterial revascularization procedure, or
  * amputation due to atherosclerotic disease.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Peripheral Artery Disease Receiving Evolocumab + High Dose Statins: Adult patients with a history of Peripheral Artery Disease (PAD) defined as one or more of the following:
  * Documented history of PAD
  * Previous limb or foot amputation for arterial vascular disease (i.e., excludes trauma),
  * Carotid artery disease (defined as >50% stenosis or prior revascularization )
  Evolocumab: Participants will be treated with high dose statins for 8 weeks followed by 8 weeks of high dose statin + evolocumab (420mg/4 wk) therapy.
Period: High Dose Statin Run-In Period (8 Weeks)
Arm/Group | Patients With Peripheral Artery Disease Receiving Evolocumab + High Dose Statins
Started | 30
Completed | 26
Not Completed | 4
Not completed — Withdrawal by Subject | 4
Period: High Dose Statins + Evolocumab (8 Weeks)
Arm/Group | Patients With Peripheral Artery Disease Receiving Evolocumab + High Dose Statins
Started | 26
Completed | 24
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Patients With Peripheral Artery Disease Receiving Evolocumab + High Dose Statins: Adult patients with a history of Peripheral Artery Disease (PAD) defined as one or more of the following:
  * Documented history of PAD
  * Previous limb or foot amputation for arterial vascular disease (i.e., excludes trauma),
  * Carotid artery disease (defined as >50% stenosis or prior revascularization )
  Evolocumab: Sixty subjects will be treated with high dose statins for 8 weeks followed by 8 weeks of high dose statin + evolocumab (420mg/4 wk) therapy.
Arm/Group | Patients With Peripheral Artery Disease Receiving Evolocumab + High Dose Statins
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Difference Between ADP-induced % Maximum Platelet Aggregation Between V2 (After 8 Weeks of HD Statin Therapy) and V5 (8 Weeks of Continued HD Statin Therapy + Evolocumab)
Description: Mean difference between 5uM ADP-induced % maximum platelet aggregation between V2 [after run-in period / 8 weeks of HD statin therapy] and V5 [end of study/ 8 weeks o]f continued HD statin therapy + evolocumab]
Time Frame: Change from week 8 (V2) to week 16 (V5)
Measure: Mean (Standard Deviation); unit: % maximum aggregation
Groups:
- Patients With Peripheral Artery Disease Receiving Evolocumab + High Dose Statins: Adult patients with a history of Peripheral Artery Disease (PAD) defined as one or more of the following:
  * Documented history of PAD
  * Previous limb or foot amputation for arterial vascular disease (i.e., excludes trauma),
  * Carotid artery disease (defined as >50% stenosis or prior revascularization )
  Patients treated with high dose statins for 8 weeks followed by 8 weeks of high dose statin + evolocumab (420mg/4 wk) therapy.
Arm/Group | Patients With Peripheral Artery Disease Receiving Evolocumab + High Dose Statins
Number analyzed (Participants) | 24
% maximum aggregation | 0.71 (10.8)

2. Secondary Outcome: Difference Between Collagen-induced Platelet Aggregation Between V2 (After 8 Weeks of HD Statin Therapy) and V5 (8 Weeks of Continued HD Statin Therapy + Evolocumab)
Description: Mean difference between 4ug Collagen-induced platelet aggregation (%) between V2 [after run-in period / 8 weeks of HD statin therapy] and V5 [end of study/ 8 weeks of continued HD statin therapy + evolocumab]
Time Frame: Change from week 8 (v2) to week 16 (v5)
Measure: Mean (Standard Deviation); unit: % maximum aggregation
Arm/Group | Patients With Peripheral Artery Disease Receiving Evolocumab + High Dose Statins
Number analyzed (Participants) | 24
% maximum aggregation | 1.4 (17.7)

3. Secondary Outcome: Difference Between SFFLRN-induced Platelet Aggregation Between V2 (After 8 Weeks of HD Statin Therapy) and V5 (8 Weeks of Continued HD Statin Therapy + Evolocumab)
Description: Mean difference between SFFLRN-induced maximum platelet aggregation (%) between V2 [after run-in period / 8 weeks of HD statin therapy] and V5 [end of study/ 8 weeks of continued HD statin therapy + evolocumab]
Time Frame: Change from week 8 (v2) to week 16 (v5)
Measure: Mean (Standard Deviation); unit: % maximum aggregation
Arm/Group | Patients With Peripheral Artery Disease Receiving Evolocumab + High Dose Statins
Number analyzed (Participants) | 24
% maximum aggregation | 6.8 (23.4)

4. Secondary Outcome: Difference Between Activated % P-selectin Positive Platelets Between V2 (After 8 Weeks of HD Statin Therapy) and V5 (8 Weeks of Continued HD Statin Therapy + Evolocumab)
Description: Mean difference in activated % P-selectin positive platelets between V2 [after run-in period / 8 weeks of HD statin therapy] and V5 [end of study/ 8 weeks o]f continued HD statin therapy + evolocumab]
Time Frame: Change from week 8 (v2) to week 16 (v5)
Population: Data not available from 3 participants due to laboratory equipment malfunction
Measure: Mean (Standard Deviation); unit: % P-Selectin Positive Platelets
Arm/Group | Patients With Peripheral Artery Disease Receiving Evolocumab + High Dose Statins
Number analyzed (Participants) | 22
% P-Selectin Positive Platelets | 126 (150)

5. Secondary Outcome: Difference in TEG MAKH Between V2 (After 8 Weeks of HD Statin Therapy) and V5 (8 Weeks of Continued HD Statin Therapy + Evolocumab)
Description: Mean difference TEG MAKH (platelet-fibrin clot strength) between V2 [after run-in period / 8 weeks of HD statin therapy] and V5 [end of study/ 8 weeks of continued HD statin therapy + evolocumab] Thromboelastography (TEG) is a viscoelastic hemostatic assay that measures the global viscoelastic properties of whole blood clot formation under low shear stress. TEG shows the interaction of platelets with the coagulation cascade (aggregation, clot strengthening, and fibrin cross-linking). MAKH is a measure of maximum platelet-fibrin clot strength. The normal range for MAKH is 53-68mm.
Time Frame: Change from week 8 (v2) to week 16 (v5)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Patients With Peripheral Artery Disease Receiving Evolocumab + High Dose Statins
Number analyzed (Participants) | 24
mm | 1.2 (3.2)

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- High Dose Statins (8 Weeks): Participants treated with high dose statins for 8 weeks
- High Dose Statins + Evolocumab (8 Weeks): Participants treated with high dose statins + evolocumab (420mg/4 wk.) for the next 8 weeks.
Arm/Group | High Dose Statins (8 Weeks) | High Dose Statins + Evolocumab (8 Weeks)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/30 | 3/26
Other Adverse Events (participants affected / at risk) | 1/30 | 5/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Statins (8 Weeks) (N=30) | High Dose Statins + Evolocumab (8 Weeks) (N=26)
Cardiac intervention (Cardiac disorders) | 0 (0) | 3 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Statins (8 Weeks) (N=30) | High Dose Statins + Evolocumab (8 Weeks) (N=26)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Allergic Rhinitis (Immune system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Elevated Liver Enzymes (Hepatobiliary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT03247972/Prot_SAP_000.pdf